CLINICAL TRIAL: NCT04083456
Title: Improving Health Self-Management Using Walking Biobehavioral Intervention for People With Dysvascular Lower Limb Amputation
Brief Title: Dysvascular Amputation Self-Management of Health
Acronym: DASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-0534; R01NR018450 (NIH)
Record Dates: First submitted 2019-08-19; First posted 2019-09-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Amputation; Diabetes Mellitus; Peripheral Artery Disease
Keywords: Amputation; Dysvascular Amputation; Diabetes; Peripheral Artery Disease; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled futility design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Biobehavioral Intervention (EXP) (Experimental): The EXP group will receive biobehavioral training that is integrated into the conventional outpatient training component and is delivered over 5 months. There will be 10 biobehavioral sessions, 1 of which will be a combined biobehavioral/conventional outpatient session and the other 9 being telehealth sessions.
  Interventions: Behavioral: Walking Biobehavioral Intervention
- Attention Control (CTL) (Active Comparator): The CTL group intervention will include the same conventional outpatient training (10 sessions) as the EXP group and receive the same computer tablets with telehealth software as the EXP group (week 3 of prosthetic training).
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Walking Biobehavioral Intervention — Each walking biobehavioral training session includes self-monitoring, tailored feedback, identification of barriers and facilitators, problem solving, action planning and encouragement. Self-monitoring of walking behavior will occur with participant use of the FitBit sensor and software, reviewed with the interventionist at each session. Tailored feedback from the FitBit sensor, as well as feedback from the interventionist, will detail progress over time and be compared to baseline data. Barriers and facilitators of reaching activity goals will be discussed with emphasis on problem solving to take advantage of facilitators and minimize/remove participant-specific barriers. Action planning will be based on weekly step goals set collaboratively by the interventionist and participant, based the FitBit data. Finally, encouragement will be provided by the interventionist by putting progress or lack of progress in perspective of the efforts made by the participant.
  Arms: Walking Biobehavioral Intervention (EXP)
Other: Attention Control — Attention control sessions will include a brief review of the conventional home-exercises, a summary of all healthcare visits and falls, and interventionist-delivered education on safety topics (e.g., fall prevention, wound care, assistive device use). Outpatient therapists will provide home-based exercises to ensure that the participant receives adequate training and demonstrates safe performance prior to home use. The CTL interventionist will assess and discuss the safe performance of each home-based exercise with CTL group participants. Exercises in the CTL group will only be progressed by the outpatient physical therapist and not during the telehealth sessions.
  Arms: Attention Control (CTL)

SUMMARY:
The purpose of this study is to determine if walking biobehavioral intervention improves physical activity after dysvascular lower limb amputation.

DETAILED DESCRIPTION:
Sedentary lifestyles and high levels of disability are relevant public and personal health issues resulting from the chronic comorbid condition of dysvascular lower limb amputation. This study examines the use of an evidence-based walking biobehavioral intervention to increase physical activity after dysvascular amputation. The proposed intervention leverages successes in conventional prosthetic rehabilitation, while addressing the complex health conditions and chronic sedentary behaviors that underlie dysvascular amputation, with the ultimate goal of improved physical activity self-management to minimize disability.

ELIGIBILITY:
Inclusion Criteria:

* Within the age range of 50-85 years
* Confirmed diagnosis of Type II Diabetes Mellitus (DM) and/or Peripheral Artery Disease (PAD)
* Transtibial, knee disarticulation, or transfemoral lower-limb amputation (LLA) (or re-amputation) within the past 12 months
* Participant goal of household walking or better using a prosthesis

Exclusion Criteria:

* Trauma or cancer-related etiology of the LLA
* Decisionally challenged individuals (MMSE score below 24)
* Prisoners
* Active cancer treatment
* Recent stroke (within 2 years)
* Clinical discretion of principal investigator to exclude patients who are determined to be unsafe and/or inappropriate to participate in the described intervention.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Day 0 (start of conventional prosthetic rehabilitation), prosthetic rehabilitation end (3 months), intervention end (6 months), and 6 months after intervention end (12 months)
  Change in 10 day physical activity step count with ActivPAL activity monitor between the beginning of conventional prosthetic rehabilitation to the end of intervention. Maintenance will be observed at six months after the end of the intervention.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS): Self-Efficacy for Managing Symptoms | Day 0, 3 months, 6 months and 12 months
  Change in participant's confidence in managing symptoms of chronic disease. Final scores range from 4 points (not at all confident) to 20 points (very confident).
PROMIS: Self-Efficacy for Managing Daily Activities | Day 0, 3 months, 6 months and 12 months
  Change in participant's confidence in managing daily activities. Final scores range from 4 points (not at all confident) to 20 points (very confident).
PROMIS: Ability to participate in social roles and activities | Day 0, 3 months, 6 months and 12 months
  Change in participant's ability to participate in social roles and activities. Final scores range from 8 points (never participates) to 40 points (always participates).
Prosthesis Evaluation Questionnaire - Mobility Score | Day 0, 3 months, 6 months and 12 months
  Change in self-reported mobility. Final scores range from 0 (lowest mobility) to 4 (highest mobility)
Timed Up-and-Go test | Day 0, 3 months, 6 months and 12 months
  Change in time required to rise from chair, walk 10 feet, turn around and return to sitting in same chair.
World Health Organization-Disability Assessment Schedule 2.0 | Day 0, 3 months, 6 months and 12 months
  Change in self-reported disability. Final scores range from 0 (no disability) to 100 (full disability).
Self-Efficacy for Managing Chronic Disease | Day 0, 3 months, 6 months and 12 months
  Change in self-reported confidence in managing different aspects of chronic disease. Final scores range from 1 (not at all confident in managing chronic disease) to 10 (totally confident in managing chronic disease).

OTHER OUTCOMES:
Activities-specific Balance Confidence Scale | Day 0, 3 months, 6 months and 12 months
  Change in self-reported balance confidence. Final scores range from 0% (no confidence in balance) to 100% (complete confidence in balance).
Two-Minute Walk Test | Day 0, 3 months, 6 months and 12 months
  Change in the distance a participant can walk in two minutes. Use of assistive device is noted
Five Meter Walk | Day 0, 3 months, 6 months and 12 months
  Change in the length of time it takes a participant to walk 5 meters, at a comfortable walking pace.
Study Intervention Reach | Day 0
  Percentage of eligible participants enrolled
Outpatient Practitioner Intervention Fidelity | Day 0 through 3 months
  An individual practitioner's percent adherence to outpatient intervention protocol
Biobehavioral Practitioner Intervention Fidelity | Day 0 through 6 months
  An individual interventionist's percent adherence to biobehavioral intervention protocol
FitBit Use Adherence | Month 12
  Number of days participant uses FitBit during the no-contact phase of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cory Christiansen, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish the trial results data on the ClinicalTrials.gov website, on which the clinical trial will be registered. Sharing of data will include the potential of sharing raw data generated from all clinical assessments under a data-sharing agreement.
Supporting Information: ICF, CSR
Time Frame: The investigators will publish the trial results within one year of testing the final participant.
Access Criteria: User registration will be required to access/download any data and will require agreement to conditions of use in accordance with NIH Data Sharing Policy Guidelines.

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273